CLINICAL TRIAL: NCT01021826
Title: Determinants of Perioperative Hyperglycaemia in Primary Hip and Knee Replacement
Brief Title: Perioperative Hyperglycaemia in Primary Total Hip and Knee Replacement
Acronym: HyTe-1
Status: Completed | Type: Observational
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Esa Jamsen, MD, PhD, Researcher, Coxa, Hospital for Joint Replacement
Other Study IDs: HyTe-1
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Knee Replacement; Hip Replacement; Hyperglycemia
Keywords: knee replacement; hip replacement; hyperglycemia; diabetes; osteoarthritis
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma sample (one per patient, collected before surgery)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip and knee replacements recipients: Osteoarthritis patients undergoing elective primary hip and knee replacement and being followed-up in this study.

SUMMARY:
The purpose of this study is to analyze how common stress hyperglycaemia (abnormally high blood glucose) is in primary hip and knee replacement surgeries and which factors predispose to hyperglycaemia.

DETAILED DESCRIPTION:
Postoperative infections remain one of the most frequent reasons of failure of hip and knee prostheses. Diabetes increases the risk of infections. In other fields of surgery, hyperglycemia induced by surgical stress (stress/perioperative hyperglycemia) has been associated with higher rates of postoperative infections and complications. Such studies have not yet been performed in the field of joint replacement surgery. Unlike several other risk factors of infected joint replacements, hyperglycemia is potentially modifiable and therefore its prevalence, predisposing factors and association with postoperative infections are of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis
* Scheduled for primary hip or knee replacement

Exclusion Criteria:

* Arthritis other than osteoarthritis
* Medication affecting glucose metabolism (excl. antidiabetic agents)
* Not undergoing hip or knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Occurrence (and severity) of hyperglycemia following primary hip or knee replacement | 3 days (average)
  Follow-up covers postoperative hospital stay at the operating hospital, that lasts typically 2-5 days.

SECONDARY OUTCOMES:
Incidence of surgical-site infections | 1 year
Prevalence of glucose metabolism disorders and metabolic syndrome | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Moilanen, MD, PhD, Study Director — Coxa, Hospital for Joint Replacement; Esa Jämsen, MD, PhD, Principal Investigator — Coxa, Hospital for Joint Replacement; Pasi Nevalainen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Coxa, Hospital for Joint Replacement, Tampere, Finland

REFERENCES:
- [Result] Jamsen E, Nevalainen PI, Eskelinen A, Kalliovalkama J, Moilanen T. Risk factors for perioperative hyperglycemia in primary hip and knee replacements. Acta Orthop. 2015 Apr;86(2):175-82. doi: 10.3109/17453674.2014.987064. Epub 2014 Nov 18. PMID 25409255